CLINICAL TRIAL: NCT06880757
Title: 177Lu-FAP-2286 Treatment in Urethelial Neoplasms: Utility and Safety as a Novel Treatment.
Acronym: FAUNUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Cigdem Soydal, Prof of Nuclear Medicine, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KAEK-05
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer Metastatic or Unresectable
Keywords: Bladder Cancer; Radionuclide treatment; Dosimetry
MeSH Terms: conditions — Neoplasm Metastasis; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients with metastatic bladder cancer who will received Lu-177 FAPI treatment
  Interventions: Other: Radionuclide treatment with Lu-177 FAPI

INTERVENTIONS:
Other: Radionuclide treatment with Lu-177 FAPI — Systemic radionuclide treatment with Lu-177 FAPI

SUMMARY:
Ga-68-FAPI has recently been proven to be superior to F-18-FDG in various cancers. These results have also raised hope in using FAP radiopharmaceuticals with theranostic approach. Lu-177 bound FAPI molecules have been started to be used in some cancers in clinical trials following its efficacy proven by case reports. Similarly,as a pilot study, this project aims to investigate safety and efficacy of Lu-177- FAP-2286 in metastatic urothelial carcinomas of bladder.

A total of 10 histopathologically proven urothelial bladder cancer patients >18y of age will be included in the study. After taking informed consent, all patients will undergo both 18F-FDG PET/CT and 68Ga-FAPI PET/CT for restaging before initiation of Lu-177-FAP-2286. Patients who show progression despite advanced therapies and high Ga-68 FAPI uptake will be enrolled. Patients with histopathologically proven advanced stage urothelial bladder cancer refractory to all standard therapies and no standard treatments are available or are contraindicated. Radiopharmaceutical will be administered 150mCi fixed dose, 3 cycles, 8 weeks interval. Posttherapy whole body SPECT/CT imaging will be obtained 4.,24.,96,120Hours of treatment for dosimetric calculations. All patients will be monitored for safety issues and possible long term side effects. Hematological tests, renal and liver function tests will be performed every 2 weeks, radiological imaging for tumor response assessment will be performed every 6 weeks. Symptoms will be taken under consideration for symptomatic response QoL questioner. In case of objective progression, therapy will be stopped. Otherwise, will be completed to 4 cycles.

Administration of Lu-177 FAPİ treatment will be performed by 1st partner from Turkey. Posttreatment SPECT/CT images will be obtained and collected for dosimetric calculations. Heatly organ doses and tumor doses will be calculated bt 2nd partner form Italy in collaboration with 1st partner. In consideration of the advances in radionuclide treatments to achieve objective response within safety margins to healthy organs, dosimetric approaches are mandatory. As a novel treatment dosimetric data for Lu-177 FAPİ treatment is limited. Despite to being a reference center for radionuclide treatments 1st partner has no experience on dosimetric calculations for systemic radionuclide treatments. As an experienced center for dosimetric studies, 2nd partner will be a milestone for analysis of dose response and toxicity analyses for this pilot study of novel treatment.

DETAILED DESCRIPTION:
Bladder cancer has a variable incidence worldwide, changing with environmental factors. Urothelial carcinoma the the most common histopathological subtype. Early-stage bladder cancer has a favoruable prognosis, despite high survival rates (5years survival rate 40-70%). Advanced stage, however, has a very poor prognosis, with high metastatic rate. In these patients, several agents have been tried to improve outcomes. Radionuclide therapies gained importance in multiple cancer types, including prostate carcinoma, with recent reports proving its efficacy in especially metastatic, inoperable, advanced stage disease (1-4). In advanced stage bladder cancer, the role of radionuclide treatments has not been investigated yet. But in case a metabolic pathway can be viualised by a diagnostic radiopharmaceutical, then radiolabeled lesions can also be cured by the theranostic pair. Although F-18-FDG is a very good agent for detecting metastatic disease in bladder cancer, it cannot be used for theranostic purposes. Other routes are thus investigated for this aim.

Fibroblast activation protein (FAP) is highly expressed in the stroma of several tumor entities. Especially breast, colon, and pancreatic carcinomas are characterized by a strong desmoplastic reaction, which means that 90% of the gross tumor mass can consist of stromal but not tumor cells. Fibroblasts are present ubiquitously in the whole body and show very low or no FAP expression. In contrast, cancer-associated fibroblasts are specifically characterized by the expression of FAP (5).

Thus, cancer-associated fibroblasts differ from normal fibroblasts by providing FAP as a target with a relatively high tumor-specific expression, and FAP inhibitors (FAPIs) have already been developed as cancer drugs (6,7). Based on a quinoline-based FAP-specific inhibitor (6), a new class of radiopharmaceuticals was designed and found preclinically highly promising as molecular targeting imaging probes, and it is hoped that they also will be therapeutically useful (8,9).

First-in-human cases demonstrated high-contrast tumor imaging in various cancers, including bladder cancer (8-11). Thus, it has also been recognized as a promising target for therapy. To date, there are no studies available investigating FAPI targeted radionuclide therapy in bladder cancer.

The major aim of this study is investigating the safety and efficacy of Lu-177 FAP-2286 in advanced stage urothelial bladder cancer. The study is planned as a pilot study in a relatively small group of patients.

For non-standardised therapies, radionuclide therapies are adviced to be given with a dosimetric approach. In personalized therapies, dosimetry allows improved safety and efficacy, easier monitorisation of therapy, accurate measurement of radiation doses and thus minimizing adverse event rates while maximizing the therapeutic benefit in the targeted areas. So the secondary aim of this study is to make a dosimetric study, including the investigation of physiological distribution and pharmacokinetics-pharmacodynamics of this novel radiopharmaceutical.

Proving safety and efficacy in this pilot study will lead to open a window for its use in further clinical studies conducted in larger patient populations. Supported by further studies, a new therapeutic option will hopefully be developed for incurable bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically proven advanced stage urothelial bladder cancer refractory to all standard therapies and no standard treatments are available or are contraindicated.

  * Patients aged >18y, male or female gender
  * Patients who are willing to cooperate with the study protocol, including the therapy regimen, posttherapy imaging and follow up visits
  * Patients who read and signed the written informed consent form.
  * A positive Ga-68-FAPI scan result (at least 50% of the lesions with an SUVmax >1.5 times liver SUVmax )
  * Blood tests (Platelets>120.000/mm3, Neutrophils>1500cell/mm3, Hb>8g/dL
  * Liver function tests: (ALT and AST<2.5Xupper limit of normal, Bilirubin<2mg/dL, Total bilirubin<1.5X upper limit of normal
  * PT, aPTT and INR in normal range
  * Normal GFR, serum Cr levels
  * ECOG 0-1
  * Life expectancy longer than 6 months

Exclusion Criteria:

* Low Ga-68-FAPI uptake
* Not willing to sign informed consent form
* ECOG >1
* Hematological tests and renal function tests are not eligible
* Disseminated bone marrow metastasis
* Central nervous system metastasis or existence of any lesion with risk of compression
* Co-existing secondary malignancies
* Previous radioligand therapies
* Being received anticancer therapies in 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Lu-177-FAP-2286 | 1 to 30 months
  Efficacy of Lu-177-FAP-2286 based on objective response rate according to RECIST.
Dosimetry of Lu-177-Fap-2286 | 6 to 30 months
  Radiation dosimetry of Lu-177-FAP-2286 to tumoral lesions and healthy organs measured by absorbed dose estimates (Gy)
Safety of Lu-177-FAP-2286 | 6 to 36 months
  Determination of short and long term adverse events

IPD SHARING:
Plan to Share IPD: Undecided